CLINICAL TRIAL: NCT06174116
Title: Metabolic Effects of Adjunctive Lumateperone Treatment in Clozapine-Treated Patients With Schizophrenia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Principal Investigator, Xiaoduo Fan, MD, MPH, Director, UMass Mind, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001339
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: Clozapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — lumateperone

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 Placebo capsules taken orally per day for 12 weeks
  Interventions: Drug: Placebo
- Lumateperone (Experimental): 42mg (two 21mg capsules) lumateperone (Caplyta) taken orally per day for 12 weeks
  Interventions: Drug: Lumateperone

INTERVENTIONS:
Drug: Lumateperone — Subject will take lumateperone (Caplyta) for 12 weeks, in addition to their regular medications.
  Other Names: Caplyta
  Arms: Lumateperone
Drug: Placebo — Subject will take placebo for 12 weeks, in addition to their regular medications.
  Arms: Placebo

SUMMARY:
The main question this study is trying to answer is whether lumateperone, an FDA-approved antipsychotic drug, can help reduce possible side effects of clozapine, such as weight gain and elevated levels of sugar and bad cholesterol.

Participants will be randomly assigned to either take lumateperone (Caplyta) or a placebo for 12 weeks, in addition to their regularly prescribed clozapine. During their participation, patients will answer questions about their psychiatric and daily functioning, have blood drawn, and have their body composition analyzed (similar to stepping on a scale).

DETAILED DESCRIPTION:
This is a 12-week study in which we investigate how adjunctive lumateperone affects lipid particle size and body composition in clozapine-treated patients with schizophrenia; in addition, we will investigate if lumateperone improves insomnia. Outcome measures will record a variety of assessments related to participants' psychiatric symptoms, psychosocial functioning, and biological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-5 criteria for diagnoses of schizophrenia or schizoaffective disorder based on the MINI International Neuropsychiatric Interview (MINI 7.0)
* On clozapine treatment for at least 6 months
* Stable dose of antipsychotic treatment for at least 1 month
* Well established compliance with outpatient medications
* Subjects of child-bearing potential are required to practice appropriate birth control methods during the study.

Exclusion Criteria:

* Psychiatrically unstable per clinical judgement by the principal investigator
* Patients not on stable dose of antipsychotic medications
* Currently meets DSM-5 criteria for any substance use disorder other than caffeine and nicotine
* Significant, unstable medical conditions including severe cardiovascular, hepatic, renal or other medical diseases
* History of a seizure disorder
* Pregnancy or breastfeeding
* On lumateperone treatment in the past 3 months
* On a dopamine partial agonist antipsychotic agent in the past 3 months (aripiprazole, brexpiprazole, cariprazine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Week 0, Week 6, and Week 12
  Participant Body Mass Index will be measured by standard methods
Waist Circumference | Week 0, Week 6, and Week 12
  Participant Waist Circumference will be measured by standard methods
Body Composition - Fat Mass | Week 0 and Week 12
  Body Composition will be assessed using the research-grade medical body composition analyzer Seca 515/514. Fat mass will be measured in grams.
Body Composition - Total Body Mass | Week 0 and Week 12
  Body Composition will be assessed using the research-grade medical body composition analyzer Seca 515/514. Total Body Mass will be measured in grams.
Body Composition - Fat Percentage | Week 0 and Week 12
  Body Composition will be assessed using the research-grade medical body composition analyzer Seca 515/514. Fat Percentage will be calculated as fat mass (in grams) divided by total mass (in grams).
HBA1C | Week 0 and Week 12
  Participant HBA1C will be measured using standard labs
Fasting Insulin | Week 0, Week 6, and Week 12
  Participant Fasting Insulin will be measured using standard labs
LDL Particle | Week 0 and Week 12
  LDL particle size will be determined using the NMR spectroscopy (LipoScience, Raleigh, NC)
Small LDL Particle | Week 0 and Week 12
  Small LDL particle size will be determined using the NMR spectroscopy (LipoScience, Raleigh, NC)
Large HDL Particle | Week 0 and Week 12
  Large HDL Particle size will be determined using the NMR spectroscopy (LipoScience, Raleigh, NC)
Large VLDL Particle | Week 0 and Week 12
  Large VLDL Particle size will be determined using the NMR spectroscopy (LipoScience, Raleigh, NC)

SECONDARY OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) | Week 0, Week 6, and Week 12
  PANSS is a measure used to assess symptom severity in patients with schizophrenia. It consists of three sections: Positive scale has 7 items, Negative scale has 7 items, and General Psychopathology has 16 items. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme.
Calgary Depression Scale (CDRS) | Week 0, Week 6, and Week 12
  The CDRS is used to assess depression symptoms in patients with schizophrenia.
Clinical Global Impression - Severity Scale (CGI-S) | Week 0, Week 6, and Week 12
  The CGI-S is an observer rated scale. The CGI-S measures illness severity on a 7-point Likert scale 1) Normal, not at all ill, 2) Borderline mentally ill, 3) Mildly ill, 4) Moderately ill, 5) Markedly ill, 6) Severely ill, and 7) Among the most extremely ill patient.
Clinical Global Impression - Improvement Scale (CGI-I) | Week 0, Week 6, and Week 12
  The CGI-I is an observer rated scale. The CGI-I is used to measure improvement in illness and uses a 7-point Likert scale: 1) Very much improved, 2) Much improved, 3) Minimally improved, 4) No change 5) Minimally worse, 6) Much worse, 7) Very much worse.
Insomnia Severity Index (ISI) | Week 0, Week 6, and Week 12
  The ISI is a 7-question survey assessing symptoms of insomnia. The maximum score is 28 with higher scores indicating greater severity. The ISI is a reliable and valid instrument to assess insomnia and treatment response.
Henrichs Carpenter Quality of Life Scale (QLS) | Week 0, Week 6, and Week 12
  The QLS is a 21-item scale providing information on symptoms and functioning in patients with schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No